CLINICAL TRIAL: NCT06563557
Title: ERASME ULB: Erasme Randomized Controlled Trial Surveys Hemodynamic Excursions During Esophagectomy - a Double Blind Study
Brief Title: Erasme Randomized Controlled Trial Surveys Hemodynamic Excursions During Esophagectomy
Acronym: ERASME ULB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: P2023/514 /B4062024000032
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-06

CONDITIONS: Esophagectomy; Epidural; Anesthesia; Paravertebral Anesthesia; Hemodynamic Instability

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural group (Active Comparator)
  Interventions: Other: Hemodynamic changes between epidural and paravertebral during esophagectomy
- Paravertebral group (Experimental)
  Interventions: Other: Hemodynamic changes between epidural and paravertebral during esophagectomy

INTERVENTIONS:
Other: Hemodynamic changes between epidural and paravertebral during esophagectomy — The thoracic epidural technique remains the gold standard for perioperative pain management for this procedure. The placement of a paravertebral catheter homolateral with the thoracic incisions is strongly recommended. A goal directed fluid therapy is proposed to guide fluid management and limit postoperative complications. Few studies suggested less side effects in the paravertebral group. The vasoplegia due to the epidural can cause significant hypotension especially as reverse Trendelenburg position is required during surgery. The aim is to bring more light to the hemodynamic changes caused by two different locoregional techniques. An algorithm for fluid and vasopressor management has been proposed. We defined hypotension as 20% of decrement of the median arterial pressure during anesthesia. To reduce bias, the locoregional techniques is performed by an experienced anesthesiologists and the rest of the perioperative management is conducted by another blinded anesthesiologist.

SUMMARY:
In our high volume center, the majority of esophagectomy procedures are performed with minimally invasive techniques. The thoracic epidural technique remains the gold standard and homolateral paravertebral catheter is strongly recommended. The vasoplegia and sympathetic blockade due to the epidural can cause significant hypotension especially as reverse Trendelenburg position is required during surgery. The aim is to study hemodynamic changes caused by two different techniques. Previous studies found a similar pain management between both locoregional techniques, however few studies suggested less side effects in the paravertebral group during major abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Adult, Capable of giving consent, two or three incisions esophagectomy (thoracoscopic/ thoracotomy) no laparotomy

Exclusion Criteria:

* patient refusal, total language barrier, coagulation disorders, thrombocytopenia <75 000, contraindications to locoregional anesthesia (infection local site, allergy to local anesthesic), scoliosis Cobb > 45%, atrial fibrillation, end stage renal disease),

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Consumption of norepinephrine and fluids during procedure | 6 hours
  norepinephrine mcg/kg/hr

SECONDARY OUTCOMES:
Postoperative complications | 6 months
  Medical complications: Pneumonia, atrial fibrillation, thromboembolic event Surgical complications : Wound dehiscence, anastomotic leakage, chylothorax, recurrent laryngeal nerve injury

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo SZEGEDI, PHD, Study Chair — Laszlo.szegedi@hubruxelles.be

REFERENCES:
- [Background] Low DE, Allum W, De Manzoni G, Ferri L, Immanuel A, Kuppusamy M, Law S, Lindblad M, Maynard N, Neal J, Pramesh CS, Scott M, Mark Smithers B, Addor V, Ljungqvist O. Guidelines for Perioperative Care in Esophagectomy: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations. World J Surg. 2019 Feb;43(2):299-330. doi: 10.1007/s00268-018-4786-4. PMID 30276441
- [Background] Deana C, Vetrugno L, Bignami E, Bassi F. Peri-operative approach to esophagectomy: a narrative review from the anesthesiological standpoint. J Thorac Dis. 2021 Oct;13(10):6037-6051. doi: 10.21037/jtd-21-940. PMID 34795950
- [Background] Kingma BF, Eshuis WJ, de Groot EM, Feenstra ML, Ruurda JP, Gisbertz SS, Ten Hoope W, Marsman M, Hermanides J, Hollmann MW, Kalkman CJ, Luyer MDP, Nieuwenhuijzen GAP, Scholten HJ, Buise M, van Det MJ, Kouwenhoven EA, van der Meer F, Frederix GWJ, Cheong E, Al Naimi K, van Berge Henegouwen MI, van Hillegersberg R. Paravertebral catheter versus EPidural analgesia in Minimally invasive Esophageal resectioN: a randomized controlled multicenter trial (PEPMEN trial). BMC Cancer. 2020 Feb 22;20(1):142. doi: 10.1186/s12885-020-6585-1. PMID 32087686
- [Background] van den Berg JW, Tabrett K, Cheong E. Paravertebral catheter analgesia for minimally invasive Ivor Lewis oesophagectomy. J Thorac Dis. 2019 Apr;11(Suppl 5):S786-S793. doi: 10.21037/jtd.2019.03.47. PMID 31080659
- [Background] Yeung JH, Gates S, Naidu BV, Wilson MJ, Gao Smith F. Paravertebral block versus thoracic epidural for patients undergoing thoracotomy. Cochrane Database Syst Rev. 2016 Feb 21;2(2):CD009121. doi: 10.1002/14651858.CD009121.pub2. PMID 26897642